CLINICAL TRIAL: NCT00249834
Title: A Phase IIIB/IV, Open Label Study to Assess the Efficacy and Safety of a Pre-defined, Fixed Dose of Gonal-f® (Filled-by-Mass in a Prefilled Pen) Based on Subject Baseline Characteristics, for Ovarian Stimulation in Subjects Undergoing in Vitro Fertilization (IVF)
Brief Title: Safety and Efficacy of Pre-defined, Fixed Dose of Gonal-f Pen Based on Subject Baseline Characteristics in Subjects Undergoing in Vitro Fertilization (IVF)
Acronym: CONSORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25198
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2017-08

CONDITIONS: Infertility
Keywords: Assisted Reproductive Technology (ART); Infertility; Ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit; Chorionic Gonadotropin

ARMS (8):
- Gonal-f 112.5 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 37.5 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 75 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 150 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 187.5 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 225 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 262.5 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)
- Gonal-f 300 IU (Experimental)
  Interventions: Drug: Gonal-f; Drug: Recombinant human chorionic gonadotrophin (r-hCG)

INTERVENTIONS:
Drug: Gonal-f — GONAL-f (follitropin alfa) will be administered subcutaneously based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle.
  Other Names: follitropin alfa; Recombinant Human Follicle Stimulating Hormone (r-hFSH)
Drug: Recombinant human chorionic gonadotrophin (r-hCG) — When at least 1 follicle greater than or equal to (>=) 18 millimeter (mm) and 2 follicles >=16 mm in diameter develop, 250 microgram (mcg) of recombinant human chorionic gonadotrophin (r-hCG) will be administered.

SUMMARY:
Clinical validation of the assisted reproductive technology (ART) treatment guidelines, which determine the optimal dose of recombinant human follicle stimulating hormone (r-hFSH) based on subject baseline characteristics/predictors of ovarian response.

ELIGIBILITY:
Inclusion Criteria

* Be an infertile subject justifying an in-vitro fertilization/embryo transfer (IVF/ET) treatment.
* Have a male partner with semen analysis within the past six months prior to study entry considered adequate to proceed with regular insemination or intracytoplasmic sperm injection (ICSI) according to the center's standard practice. If these criteria are not met, the subject can only be entered if donor sperm will be used.
* Be between her 18th and 35th birthday (35 not included).
* Have a regular spontaneous ovulatory menstrual cycle between 21 and 35 days in length.
* Have early follicular phase (Day 2-4) serum levels within the last 3 months prior to study entry of:
* Follicle stimulating hormone (FSH) greater than or equal to (>=) 12 International units per liter (IU/L), and
* Oestradiol (E2) within center's local normal laboratory range values.
* Presence of both ovaries.
* Have a uterine cavity without abnormalities, which, in the investigator's opinion, could impair embryo implantation or pregnancy evolution as assessed within the last 3 years using ultrasound (US), hysteroscopy (HSC), or hysterosalpingography (HSG).
* Have a negative cervical papanicolaou (PAP) test within the last 6 months prior to study entry.
* Have at least one wash-out cycle (defined as >= 30 days since the last dose of clomiphene citrate or gonadotrophin treatment) since the last ART cycle and/or clomiphene citrate or gonadotrophin treatment prior to starting gonadotrophin releasing hormone (GnRH) agonist therapy.
* Have a negative pregnancy test prior to beginning GnRH agonist therapy.
* Be willing and able to comply with the protocol for the duration of the study. Have given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to her future medical care.

Exclusion Criteria:

* Had 2 previous ART cycles with a poor response to gonadotrophin stimulation, defined as less than or equal to (<=) 5 mature follicles and/or <=3 oocytes collected in any previous IVF cycle or hyper response, defined as >=25 oocytes retrieved.
* Any medical condition, which in the judgement of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug. In case of doubt, the subject in question should be discussed with Serono's Therapeutic Director.
* Had previous severe ovarian hyperstimulation syndrome (OHSS).
* A body mass index (BMI) greater than (>) 30 kilogram per square meter (kg/m^2)
* Any contraindication to being pregnant and/or carrying a pregnancy to term.
* Extra-uterine pregnancy within the last 3 months.
* History of 3 or more miscarriages (early or late miscarriages) due to any cause.
* Tumours of the hypothalamus and pituitary gland.
* Ovarian enlargement or cyst of unknown aetiology.
* Ovarian, uterine or mammary cancer.
* A clinically significant systemic disease.
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus.
* Abnormal gynaecological bleeding of undetermined origin.
* Known allergy or hypersensitivity to human gonadotrophin preparations.
* Any active substance abuse or history of drug, medication or alcohol abuse in the past 5 years.
* Entered previously into this study or simultaneous participation in another clinical trial

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2004-09-22 (Actual); Primary Completion 2006-01-16 (Actual); Study Completion 2006-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Medical Information, Paris, France

REFERENCES:
- [Background] Olivennes F, Howles CM, Borini A, Germond M, Trew G, Wikland M, Zegers-Hochschild F, Saunders H, Alam V; CONSORT study group. Individualizing FSH dose for assisted reproduction using a novel algorithm: the CONSORT study. Reprod Biomed Online. 2009 Feb;18(2):195-204. doi: 10.1016/s1472-6483(10)60256-8. PMID 19192339
- [Result] Olivennes F, Howies CM, Borini A, Germond M, Trew G, Wikland M, Zegers-Hochschild F, Saunders H, Alam V. Individualizing FSH dose for assisted reproduction using a novel algorithm: the CONSORT study. Reprod Biomed Online. 2011 Feb;22 Suppl 1:S73-82. doi: 10.1016/S1472-6483(11)60012-6. PMID 21575853
- See also: Full FDA approved prescribing information can be found here — http://www.fertilitylifelines.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 166 subjects received at least 1 dose of recombinant human follicle stimulating hormone (r-hFSH). Of these, 161 subjects received r-hFSH in a dose group of 5 or more subjects. As per statistical analysis plan, only dose groups having 5 or more subjects were to be analyzed for efficacy and safety analysis in this study.
Groups:
- Gonal-f 37.5 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 37.5 International Units (IU) per day based on assisted reproductive technology (ART) treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle greater than or equal to (>=) 18 millimeter (mm) and 2 follicles >=16 mm in diameter were developed, a single injection of 250 microgram (mcg) of recombinant human chorionic gonadotrophin (r-hCG) was administered.
- Gonal-f 75 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 75 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Gonal-f 112.5 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 112.5 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Gonal-f 150 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 150 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Gonal-f 187.5 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 187.5 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Gonal-f 225 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 225 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Gonal-f 262.5 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 262.5 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Gonal-f 300 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 300 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
Period: Overall Study
Arm/Group | Gonal-f 37.5 IU | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU | Gonal-f 262.5 IU | Gonal-f 300 IU
Started | 1 | 48 | 45 | 34 | 24 | 10 | 2 | 2
Completed | 0 | 29 | 31 | 26 | 19 | 8 | 1 | 2
Not Completed | 1 | 19 | 14 | 8 | 5 | 2 | 1 | 0
Not completed — Ovarian stimulation failed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failure of down-regulation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 19 | 14 | 8 | 5 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gonal-f 37.5 IU: GONAL-f (follitropin alfa) administered subcutaneously, at a dose of 37.5 IU/day based on ART treatment guidelines, which determined the optimal dose of r-hFSH based on subject baseline characteristics/predictors of ovarian response throughout stimulation cycle. When at least 1 follicle >=18 mm and 2 follicles >=16 mm in diameter were developed, a single injection of 250 mcg of r-hCG was administered.
- Total: Total of all reporting groups
Arm/Group | Gonal-f 37.5 IU | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU | Gonal-f 262.5 IU | Gonal-f 300 IU | Total
Number analyzed (Participants) | 1 | 48 | 45 | 34 | 24 | 10 | 2 | 2 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 48 | 45 | 34 | 24 | 10 | 2 | 2 | 166
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 48 | 45 | 34 | 24 | 10 | 2 | 2 | 166
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: Mean number of oocytes retrieved on the day of ovum pick up (OPU) was calculated. Oocyte retrieval was a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body. As per statistical analysis plan, efficacy analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Time Frame: Ovum pick up day (34 to 38 hours post r-hCG administration)
Population: Intention-To-Treat (ITT) population included all 161 treated subjects who received at least 1 injection of r-hFSH, and were allocated to a dosage group that contained at least 5 subjects. Here "overall number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 34 | 39 | 31 | 22 | 9
Oocytes | 8.3 (4.5) | 9.6 (6.5) | 12.1 (6.4) | 12.7 (4.3) | 8.3 (3.8)

2. Secondary Outcome: Total Dose of Recombinant Human Follicle Stimulating Hormone (r-hFSH)
Description: As per statistical analysis plan, efficacy analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Time Frame: up to end of stimulation cycle (approximately 31 days)
Population: ITT population included all 161 treated subjects who received at least 1 injection of r-hFSH, and were allocated to a dosage group that contained at least 5 subjects.
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 48 | 45 | 34 | 24 | 10
International Units (IU) | 1102.3 (671.8) | 1287.2 (447.0) | 1632.4 (341.5) | 2043.8 (276.2) | 2572.5 (552.3)

3. Secondary Outcome: Mean Number of Ovarian Stimulation Days
Description: The mean number of stimulation days were determined based on the treatment administration information collected in the case report form. Ovarian stimulation included time from first r-hFSH injection (stimulation Day) until day on which r-hCG was administered (r-hCG day). As per statistical analysis plan, efficacy analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Time Frame: up to end of stimulation cycle (approximately 31 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 48 | 45 | 34 | 24 | 10
Days | 12.5 (4.4) | 11.0 (2.9) | 10.6 (1.8) | 11.0 (1.4) | 11.5 (2.4)

4. Secondary Outcome: Percentage of Cycles Cancelled Due to Excessive or Inadequate Response to r-hFSH
Description: as for outcome 2
Time Frame: up to end of stimulation cycle (approximately 31 days)
Population: as for outcome 2
Measure: Number; unit: Percentage of cycles
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 48 | 45 | 34 | 24 | 10
Percentage of cycles
  Excessive response | 0.0 | 0.0 | 2.9 | 0.0 | 0.0
  Inadequate response | 25.0 | 8.9 | 8.8 | 8.3 | 20.0

5. Secondary Outcome: Number of Subjects Needing Dose Adjustment
Description: Number of subjects needing increase in dose, decrease in dose or increase and decrease both in dose were reported. As per statistical analysis plan, efficacy analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Time Frame: 6 days post r-hFSH treatment
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 48 | 45 | 34 | 24 | 10
subjects
  Increase | 7 | 3 | 3 | 1 | 0
  Decrease | 0 | 0 | 1 | 2 | 1
  Increase and decrease both | 2 | 3 | 0 | 0 | 0

6. Secondary Outcome: Mean Daily Recombinant Human Follicle Stimulating Hormone (r-hFSH) Dose
Description: as for outcome 2
Time Frame: up to end of stimulation cycle (approximately 31 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/day
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 48 | 45 | 34 | 24 | 10
IU/day | 84.4 (21.6) | 114.7 (16.4) | 153.6 (12.8) | 186.5 (5.8) | 223.3 (5.3)

7. Secondary Outcome: Embryo Implantation Rate
Description: Embryo implantation rate was measured as the number of gestational sacs observed divided by the number of embryos transferred multiplied by 100. As per statistical analysis plan, efficacy analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Time Frame: 35-42 days post r-hCG administration
Population: ITT population included all 161 treated subjects who received at least 1 injection of r-hFSH, and were allocated to a dosage group that contained at least 5 subjects. Here "overall number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent sacs per embryo
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 32 | 37 | 29 | 22 | 7
Percent sacs per embryo | 36.5 (42.8) | 24.3 (35.0) | 28.2 (38.9) | 37.1 (40.5) | 11.9 (20.9)

8. Secondary Outcome: Overall Pregnancy Rate, Clinical Rate and Multiple Pregnancy Rate
Description: Overall pregnancy rate was defined as the percentage of subjects with serum beta-hCG levels greater than 10 IU/L. Clinical pregnancy rate was defined as the percentage of subjects with at least 1 ultrasound confirmed gestational sac, with or without foetal heart activity. Multiple pregnancy rate was defined as the percentage of subjects with more than 1 ultrasound confirmed gestational sac in the uterus with fetal heart activity. As per statistical analysis plan, efficacy analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Time Frame: 35-42 days post r-hCG administration
Population: as for outcome 2
Measure: Number; unit: Percentage of subjects
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Number analyzed (Participants) | 48 | 45 | 34 | 24 | 10
Percentage of subjects
  Total pregnancy | 17 | 18 | 16 | 16 | 2
  Clinical pregnancy | 15 | 14 | 12 | 12 | 2
  Multiple pregnancy | 3 | 2 | 4 | 3 | 0

ADVERSE EVENTS:
Description: As per statistical analysis plan, safety analysis were performed for only those dose groups (Gonal-f 75 IU, Gonal-f 112.5 IU, Gonal-f 150 IU, Gonal-f 187.5 IU and Gonal-f 225 IU) which included more than 5 subjects.
Arm/Group | Gonal-f 75 IU | Gonal-f 112.5 IU | Gonal-f 150 IU | Gonal-f 187.5 IU | Gonal-f 225 IU
Serious Adverse Events (participants affected / at risk) | 3/48 | 3/45 | 1/34 | 1/24 | 0/10
Other Adverse Events (participants affected / at risk) | 11/48 | 15/45 | 5/34 | 10/24 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f 75 IU (N=48) | Gonal-f 112.5 IU (N=45) | Gonal-f 150 IU (N=34) | Gonal-f 187.5 IU (N=24) | Gonal-f 225 IU (N=10)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 0
Ovarian torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f 75 IU (N=48) | Gonal-f 112.5 IU (N=45) | Gonal-f 150 IU (N=34) | Gonal-f 187.5 IU (N=24) | Gonal-f 225 IU (N=10)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 7 | 0 | 5 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Post procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Uterine operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 2 | 1 | 3 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Ovarian torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other